CLINICAL TRIAL: NCT05484856
Title: Prospective Single Centre, Open Label, Single Arm Clinical Study for Autologous Adipose Tissue Derived ADSCSs in Treatment of Patients With Osteoarthritis
Brief Title: Evaluation of Clinical Efficacy of Autologous Adipose Tissue Derived ADSCSs in Treatment of Osteoarthritis (OA)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Himanshu Bansal Foundation (Other)
Responsible Party: Principal Investigator, anupama agrawal, DR, Dr. Himanshu Bansal Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAH/CLINICALTRIAL/01/2016
Record Dates: First submitted 2022-07-30; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis, Knee
Keywords: : stromal vascular fraction (SVF), adipose derived stromal cells, adipose tissue, connective tissue, osteoarthritis, therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: This is prospective, open label, single arm clinical study that will establish the safety and efficacy of adipose derived stromal cells in patients with osteoarthritis disease. Total 140 subjects were enrolled in the study. Each subject will receive intra-articular Autologous ADSC with PRP along with standard treatment for osteoarthritis disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients with Osteoarthritis A total of 140 patients ( May 2016 to june 2020) were treated with intra articular adipose derived stromal cells (ADSC)) also known as Stromal vascualr fraction administration
  Interventions: Biological: Autologous adipose tissue derived stromal cells

INTERVENTIONS:
Biological: Autologous adipose tissue derived stromal cells — autologous adipose tissue derived stromal cells is recovered as pellet after non enzymatic processing with sonication using ultrasound . This isolation process yielded an abundant population of Adipose stromal cells(ASCs) which have multipotent differentiation potential. Immunophenotype is a CD14-, CD29+, CD31-, CD34low/+, CD45-, CD73+ and CD105+ , the SVF represents the 50-70% in volume of a lipoaspirate specimen. The SVF hosts a heterogeneous cell population (110x103 cells/ml on average) comprising mainly CD105+ mesenchymal stem cells (MSC,2-- 20%), plus a wide number of CD34+ hematopoietic cells (40%)

SUMMARY:
Osteoarthritis (OA) is a degenerative disease of great morbidity in which therapies are typically palliative and only alleviate pain Mesenchymal stem cells ,adipose derived stromal cell are possible new chondroprotective regenerative treatment modalities.

Clinical Effectiveness after administration of adipose derived stromal cells along with platelet rich plasma was investigated in 140 patients having moderate to severe knee (stage 3 and 4)

Patients were evaluated and followed up for 2 year by subjective WOMAC score,six minute walking distance ,need of rescue medication Radiographic and MRI evaluation of joint space and cartilage thickness respectively

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative disease that affects the articular cartilage over time and is accompanied by alterations to the synovium, subchondral bone, ligaments, and menisci, as well as hypertrophy of the joint capsule.

Therapies are typically palliative and only alleviate pain in a symptomatic way, failing to stop cartilage degeneration and the following breakdown of other joint structures Therefore, it is crucial for researchers to tackle the challenge of creating OA-modifying therapeutics. The potential of adult mesenchymal stem cells (MSCs) and adipose derived stromal cells fraction also known as stromal vascular fraction has recently being evaluated for chondroprotective efficacy in oa knees.

The present study was taken to evaluate Clinical Effectiveness without any doubt after administration of Non enzymatically processed adipose derived stromal cells along with platelet rich plasma in large number (140 patients) having moderate to severe knee (stage 3 and 4) with objective MRI assessment and 2 year follow up.

Methods

The selection criteria included patients 50 years of age or older with symptomatic primary osteoarthritis of the knee that was defined by daily pain for the previous three months, analgesic use at least once per week, less than 30 minutes of morning stiffness, and a WOMAC score of 75 in the target knee. Grades 3 and 4 kellergen Radiographic Grading Scale of Osteoarthritis were part of the radiographic qualifying requirements. The exclusion criteria included individuals with clinically significant systemic diseases and patients with evidence of secondary knee osteoarthritis or severe osteoarthritis (joint space width-JSW 2 mm).

The WOMAC score, developed by Western Ontario and McMaster Universities, is a commonly used indicator of patients' subjective ratings of pain, joint mobility, and physical impairment. With 5, 2, and 17 questions, respectively, it assesses three dimensions: pain, stiffness, and physical function. A minimum score is 0, highest score is 96. The maximum score for each subscale is 20, 8, or 68, correspondingly .

In order to measure the six-minute walking distance (6MWD), a 50 m distance was marked in an internal hallway, and participants were instructed to walk as far and as rapidly as they could during the course of six minutes. The whole distance was calculated and noted.

Using previously described procedures, antero-posterior radiographs of the knee joints were taken with patients standing at a distance of 1 m from the X-Ray source, with the knee completely extended. The joint space width was measured at its narrowest point (minimal JSW). According to a prior publication this trend was indicated by a JSW loss of more than 0.50 mm over the trial.

Antero-posterior radiographs of the knee joints were acquired using the previously described techniques while patients stood 1 m away from the X-Ray source with their knees fully extended. At the joint space's narrowest point, the breadth was measured (minimal JSW). This tendency was shown by a JSW loss of more than 0.50 mm during the study, in accordance with a previous publication.

Patients were instructed to take etoricoxib at a dose of no more than 90 mg BD after meals if their discomfort was intolerable. They were instructed to take 30 mg of codeine as needed if the discomfort persisted and to report the next day. Aside from any symptoms or indications that the patient reported, laboratory-based hematological and biochemical tests were also performed as part of the tolerance and safety evaluations.

A microscopic examination of the synovial fluid was performed at baseline and two years after the surgery to check for abnormal cell counts. According to the degree to which they interfered with the subject's everyday activities, adverse occurrences were classified as isolated, intermittent, or chronic. The possible causal association between the supplement and the outcome was categorized as Definite/Possible/Probable/Non-Assessable/None. The institutional committee for stem cell research and therapy gave its approval to the project. All of the patients provided written consent to participate in the trial after receiving enough information.

SVF preparation :

With the help of a 3 mm aspiration cannula and tumescent solution, about 100 ml of fat was collected from each patient's belly and put into sterile, disposable 250 ml conical centrifuge tubes. The adipose tissue underwent two PBS washes before being sonically cavitated by ultrasound at 10 mega hertz ,50 W for 30 minutes with 5-minute intervals of agitation. The SVF was then extracted as a pellet by dividing the suspension into four 50 ml centrifuge tubes and centrifuging them at 500 g for five minutes. To get rid of any remaining enzyme, the pellet was washed twice with regular saline before being resuspended in PBS. The SVF suspension was spun at 500 g for 5 min after being filtered using a 100 m cell strainer. The extra fluid was dumped. The pellet was put back together with regular saline and passed through a 40 m cell strainer. Samples were collected in order to count the number of cells, assess their vitality, and cultivate, and define the stem cells.

PRP preparation: The same donor who provided the adipose tissue's peripheral blood also provided the platelet-rich plasma. ACD Solution A was added to BD yellow top vacuum tubes with 20 ml of peripheral blood, and the tubes were centrifuged at 800 g for 10 min. To obtain a platelet pellet, the plasma fraction was collected and centrifuged at 1000 g for 5 min. After that, just 3 ml of plasma remained, which was used to resuspend the platelets.

ELIGIBILITY:
Inclusion Criteria:

Outpatients who fulfilled the clinical and radiological criteria set by the American College of Rheumatology for the diagnosis of symptomatic primary knee OA

Exclusion Criteria:

1. Evidence of secondary knee OA because of injury, inflammatory or metabolic rheumatic disease, or osteonecrosis;
2. Prior intra-articular injection of hyaluronic acid (HA), including lavage and corticosteroids within the previous three months;
3. Severe knee OA, with JSW <1 mm, or surgery required on the evaluated knee in the year
4. Patients with clinically significant systemic disease

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2020-06-27 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
changes in womac score | [Time Frame: baseline,1 month,3 months,6 months, and 1year18 months and 2 year
  WOMAC, a widely used measure to assess patients' pain, joint mobility, and physical disability evaluates three dimensions, pain, stiffness, and physical function, with 5, 2, and 17 questions, respectively. The total maximum score is 96 and minimum, 0.
  the higher the worse.
changes in cartilage thickness as assessed on 1.5 T MRI | baseline and at one year and 2 year
  Using the 1.5-T field strength with standard MRI acquisition protocols, MRI was performed of each joint individually in coronal, sagittal, and transverse planes. The maximum thickness of the cartilage at posterior,meniscal and patellar level measured at the midsagittal plane through the medial condyle was considered. The medial femoral cartilage of the affected knee was chosen for measurement

SECONDARY OUTCOMES:
changes in joint space width | baseline and at one year and 2 year
  Patients were radiographed in a weight-bearing position, joints fully extended, standing at 1 m from the X-ray source20. The width was measured at the narrowest point of the Joint (JSW) Patients were radiographed in a weight-bearing position, joints fully extended, standing at 1 m from the X-ray source20. The width was measured at the narrowest point of the Joint (JSW) Patients were radiographed in a weight-bearing position, joints fully extended, standing at 1 m from the X-ray source20. The width was measured at the narrowest point of the Joint (JSW)

CONTACTS AND LOCATIONS:
Locations (1):
- Anupam Hospital, Rudrapur, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: Yes
ALL INFORMATION AT ANY TIME
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: TO BE PUBLISHED BY MAY 2023
Access Criteria: ANYONE